CLINICAL TRIAL: NCT02941978
Title: Motivational Interviewing to Support Oral AntiCoagulation Adherence in Patients With Non-valvular Atrial Fibrillation (MISOAC-AF): A Prospective Randomized Clinical Study
Brief Title: Motivational Interviewing to Support Oral AntiCoagulation Adherence in Patients With Non-valvular Atrial Fibrillation (MISOAC-AF)
Acronym: MISOAC-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Apostolos Tzikas, MD, PhD, Interventional Cardiologist, AHEPA University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Card1
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Patient Compliance; Patient Adherence
Keywords: atrial fibrillation; oral anticoagulation; motivational intervention; adherence; treatment gaps
MeSH Terms: conditions — Patient Compliance; Atrial Fibrillation | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subject on Motivational Interview (Experimental): 1. Motivational Interview - Baseline: At hospital discharge, patients assigned to the intervention group will be contacted in person by a study physician for an interactive session and will be given an educational leaflet. Both methods will aim to educate them about the risk for stroke and the importance of adherence to OAC medication. The leaflet will also provide some basic information on how to take OAC medication (doses, food interactions, skipping doses, etc.) and will describe the main clinical manifestations of side effects.
  2. Motivational Interview - Follow-up: Patients assigned to the intervention group will be contacted via telephone for a pre-specified interview at 1 week, 2 months, 6 months and 1 year after discharge. The delegated study personnel will assess whether an intervention is required and provide specific support tailored to the needs of the patient, aiming to improve adherence to OAC.
  Interventions: Behavioral: Motivational interview
- Subject Control (Active Comparator): Patients assigned to the control group will receive usual treatment and will be contacted via telephone for a pre-specified interview at 1 year after discharge for outcome assessment.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Motivational interview — Patients assigned to the intervention group receive additional medical consultation aiming to boost optimal uptake of the anticoagulation regimen prescribed. Initially (i.e., at hospital discharge), this includes a physician-patient interactive session and provision of an educational leaflet. The leaflet is designed in a culturally and linguistically conceivable template in Greek language. It uses simple terms together with both written and pictorial materials. Patients in the intervention group will also undergo short telephonic sessions at 1 week, 2 months, 6 months and 12 months following hospital discharge
  Arms: Subject on Motivational Interview
Behavioral: Control — Patients assigned to the control group receive usual treatment, corresponding to standard practice and management of hospitalized patients with AF. For both patient-groups, the choice of OAC agent and any other background therapy is left to the discretion of the treating physician.
  Arms: Subject Control

SUMMARY:
The purpose of the study is to investigate the impact of motivational interviewing in the adherence of patients with AF to oral anticoagulation (OAC) regimens. Patients assigned to the intervention group will be interviewed and guided on the importance of adherence to OAC medication, and will be contacted at 1 week, 2 months, 6 months and 1 year after discharge for educational interactive sessions. Patients in the control group will receive usual treatment and will be contacted at 1 year after discharge.

DETAILED DESCRIPTION:
Study Purpose: To investigate the impact of motivational interviewing in the adherence of patients with AF to oral anticoagulation (OAC) regimens

Trial Design: Prospective, two-arm, single-center, randomized controlled clinical trial

Sample Size: 1000 subjects

Population: Adults with Non-valvular Atrial Fibrillation (NVAF) hospitalized in the cardiology ward for any reason who receive OAC at hospital discharge.

Intervention

1. Motivational Interview - Baseline: At hospital discharge or one day before, patients assigned to the intervention group will be contacted in person by a study physician for an interactive session and will be given an educational leaflet. Both methods will aim to educate them about the risk for stroke and the importance of adherence to OAC medication, and motivate them to adhere to their OAC treatment plan.
2. Motivational Interview - Follow-up: Patients assigned to the intervention group will be contacted via telephone for a pre-specified interview at 1 week, 2 months, 6 months and 1 year after discharge. The delegated study personnel will assess whether an intervention is required and provide specific support tailored to the needs of the patient, focusing on maintaining or improving patients' adherence to OAC

Control Patients assigned to the control group receive usual treatment, corresponding to standard practice and management of hospitalized patients with AF. Patients assigned to the control group will be contacted via telephone for a pre-specified interview at 1 year after discharge for outcome assessment.

Primary Outcome: The primary outcome is overall adherence to OAC in the year after hospitalization for any reason, reported as Proportion of Days Covered (PDC) by OAC regimens. Patients with a PDC >80% will be classified as adequately adherent.

Secondary Outcomes: The secondary outcomes include:

* The rate of persistence: the proportion of patients who are on OAC after hospital discharge and continue receiving OAC at the end of the study period.
* OAC treatment gaps: the percentage of patients who have i) continuous OAC use (no treatment gaps or gaps <7 days), ii) transient treatment gaps (7-89 days), and iii) major treatment gaps (3 months or more)
* Clinical outcomes such as death, thromboembolic event, myocardial infraction or bleeding after hospitalization.

Clinical Duration:The total study duration (concerning the primary outcome) is expected to be 3-4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Patients with comorbid non-valvular AF, defined on the basis of physician-assigned diagnoses during the hospitalization or as previously documented in the medical record, and additionally documented on an electrocardiogram or 24-h Holter monitor, if available.
3. Patients that receive OAC at hospital discharge or are eligible for OAC therapy (CHA2DS2-VASc score ≥1 for males and ≥2 for females).

Exclusion Criteria:

1. Patients unable to communicate via telephone for study interviewing
2. Patients with any medical disorder that would interfere with completion or evaluation of clinical study results
3. Patients that lived in assisted-care facilities or had terminal illness.
4. Presence of metallic valves or moderate-to-severe mitral stenosis

Anticoagulated patients on an intentionally short-term OAC prescription under physician's recommendations (i.e. lone recent AF episode) will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1140 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Adherence to OAC therapy | One year
  The primary outcome is adherence to OAC therapy between the index date (date of hospital discharge) and the end of the 1-year follow-up period, assessed as Proportion of Days Covered (PDC) by OAC regimens.

SECONDARY OUTCOMES:
OAC treatment gaps | One year
  The percentage of patients who have i) continuous OAC use (no treatment gaps or gaps <7 days), ii) transient treatment gaps (7-89 days), and iii) major treatment gaps (3 months or more)
Clinical Outcomes | Three years
  Clinical outcomes such as death, thromboembolic event, myocardial infraction or bleeding after hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Apostolos Tzikas, MD, PhD, Principal Investigator — AHEPA University Hospital
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

REFERENCES:
- [Derived] Tsiartas E, Samaras A, Papazoglou AS, Kartas A, Moysidis DV, Gemousakakis E, Kamzolas O, Bekiaridou A, Doundoulakis I, Tzikas A, Giannakoulas G. Changes in CHA2DS2-VASc score and risk of ischemic stroke among patients with atrial fibrillation. Heart Vessels. 2023 Oct;38(10):1267-1276. doi: 10.1007/s00380-023-02278-1. Epub 2023 Jun 13. PMID 37311823
- [Derived] Tsagkaris C, Papazoglou AS, Kartas A, Samaras A, Moysidis DV, Vouloagkas I, Baroutidou A, Bekiaridou A, Patsiou V, Chatzisolomou A, Panteris E, Karagiannidis E, Karvounis H, Tzikas A, Giannakoulas G. Polypharmacy and Major Adverse Events in Atrial Fibrillation. J Cardiovasc Pharmacol. 2022 Dec 1;80(6):826-831. doi: 10.1097/FJC.0000000000001339. PMID 35921643
- [Derived] Baroutidou A, Kartas A, Samaras A, Papazoglou AS, Vrana E, Moysidis DV, Akrivos E, Papanastasiou A, Vouloagkas I, Botis M, Liampas E, Karagiannidis AG, Karagiannidis E, Efthimiadis G, Karvounis H, Tzikas A, Giannakoulas G. Associations of Atrial Fibrillation Patterns With Mortality and Cardiovascular Events: Implications of the MISOAC-AF Trial. J Cardiovasc Pharmacol Ther. 2022 Jan-Dec;27:10742484211069422. doi: 10.1177/10742484211069422. PMID 35006026
- [Derived] Vrana E, Kartas A, Samaras A, Vasdeki D, Forozidou E, Liampas E, Karvounis H, Giannakoulas G, Tzikas A. Indications for percutaneous left atrial appendage occlusion in hospitalized patients with atrial fibrillation. J Cardiovasc Med (Hagerstown). 2022 Mar 1;23(3):176-182. doi: 10.2459/JCM.0000000000001226. PMID 34580251
- [Derived] Tzikas A, Samaras A, Kartas A, Vasdeki D, Fotos G, Dividis G, Paschou E, Forozidou E, Tsoukra P, Kotsi E, Goulas I, Karvounis H, Giannakoulas G. Motivational Interviewing to Support Oral AntiCoagulation adherence in patients with non-valvular Atrial Fibrillation (MISOAC-AF): a randomized clinical trial. Eur Heart J Cardiovasc Pharmacother. 2021 Apr 9;7(FI1):f63-f71. doi: 10.1093/ehjcvp/pvaa039. PMID 32339234